CLINICAL TRIAL: NCT01524406
Title: A Randomized, Double-blind, Placebo Controlled, Phase I Study to Evaluate the Safety and Tolerability of 28 Day Treatment With HPP593 Capsules in Healthy Volunteers During and After Limb Immobilization
Brief Title: Safety Study of HPP593 in Subjects During and After Limb Immobilization
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: High Point Pharmaceuticals, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HPP593-103
Record Dates: First submitted 2012-01-27; First posted 2012-02-02 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Muscle Atrophy; Hypodynamia
Keywords: Muscle Atrophy
MeSH Terms: conditions — Muscular Atrophy; Hypokinesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HPP593 (Experimental)
  Interventions: Drug: HPP593
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HPP593 — Oral, twice a day.
  Arms: HPP593
Drug: Placebo — Oral, twice a day.
  Arms: Placebo

SUMMARY:
This is a safety and tolerability study investigating the effect of HPP593 in healthy volunteers during and after limb immobilization.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking.
* Subjects must be in good health, as determined by medical history, physical examination, vital signs, electrocardiogram (ECG), and clinical test results.
* Not restricted to a wheel-chair or confined to a bed.
* Weight ≥ 50.0 kg.
* BMI between 18 and 27.5 kg/m2, inclusive, at the time of screening.

Exclusion Criteria:

* Any of the following abnormalities at Screening Visit and Baseline:

  * Fasting glucose > 110 mg/dL (Screening visit only).
  * Serum creatinine > 1.5 mg/dL. If serum creatinine is >1.5 mg/dL and creatinine clearance is >60 mL/min, the subject need not be excluded
  * Troponin I level above the upper limit of normal (ULN)
  * Liver function tests (LFTs) > 1.5x ULN
* Evidence of significant organ system dysfunction (e.g. diabetes, cardiovascular disease, cirrhosis, hypogonadism, hypo- or hyperthyroidism; hypertension)
* Any fluctuations in weight (no more than ± 2% of body weight) by subject self report in the 3 months prior to the Screening Visit.
* Has received HPP593 in a previous clinical trial.
* Smoking within 6 month prior to Day -1.
* Michigan Alcohol Screening Test score greater than 2.

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Safety Evaluation | Baseline to Day 42
  Number and severity of adverse events across trial period

SECONDARY OUTCOMES:
Change in Muscle Strength | Day 1 to Day 42
Changes on Muscle Related Biomarkers | Day 1 to Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Shulin Wang, M.D., Study Director — High Point Pharmaceuticals, LLC.
Locations (1):
- Washington University School of Medicine Division of Geriatrics and Nutritional Studies, St Louis, Missouri, United States